CLINICAL TRIAL: NCT00422435
Title: The PreCiSE Trial: CoStar™ Paclitaxel-Eluting Coronary Stent Catheter System Evaluation
Brief Title: CoStar™ Paclitaxel-Eluting Coronary Stent Catheter System Evaluation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Conor Medsystems (Industry)
Responsible Party: Christophe Dubois, M.D. Principal Investigator, UH Gasthuisberg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The PreCiSE Trial: CP-03
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Disease
Keywords: Percutaneous coronary intervention (PCI); Drug eluting stent (DES)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug eluting stent (Experimental): CoStar™ Paclitaxel-Eluting Coronary Stent with SRX catheter
  Interventions: Device: CoStar™ Paclitaxel-Eluting Coronary Stent with SRX catheter

INTERVENTIONS:
Device: CoStar™ Paclitaxel-Eluting Coronary Stent with SRX catheter — Paclitaxel-Eluting Coronary Stent

SUMMARY:
This study is designed to evaluate the performance and safety of a new catheter system.

DETAILED DESCRIPTION:
This study is designed to evaluate acute Device Success, defined as attainment of <50% residual stenosis of the target lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years of age
* Eligible for percutaneous coronary intervention
* Documented stable or unstable angina pectoris (Canadian Cardiovascular Society Classification 1, 2, 3, or 4), documented ischemia, or documented silent ischemia
* Left ventricular ejection fraction ≥25% documented within the last 6 wks
* Acceptable candidate for coronary artery bypass graft surgery
* A single de novo lesion per study subject may be treated with the study device
* Each target lesion may be composed of multiple lesions but must be completely coverable by 1 study stent
* Cumulative target lesion length per vessel ≤30 mm based on a visual estimate
* RVD ≥2.5 mm to ≤3.0 mm based on a visual estimate
* Target lesion diameter stenosis ≥50% and <100% based on a visual estimate
* Target vessel has not undergone prior revascularization within the preceding 6 months
* Target lesion must be a minimum 10 mm distance from any previously treated segment of the target vessel

Exclusion Criteria:

* Known sensitivity to cobalt chromium, paclitaxel or polymeric matrices: Translute or PLGA
* Planned treatment with any other PCI device in the target vessel(s)
* MI within 72 hours prior to the index procedure
* Patient is in cardiogenic shock
* Cerebrovascular Accident within the past 6 months
* Acute or chronic renal dysfunction (creatinine >2.0 mg/dl or >150 µmol/L)
* Contraindication to ASA or to clopidogrel
* Thrombocytopenia (platelet count <100, 000/mm3)
* Active gastrointestinal bleeding within the past three months
* Any prior true anaphylactic reaction to contrast agents
* Patient is currently, or has been treated with paclitaxel (systemic) within 12 months of the index procedure
* Female of childbearing potential with a positive pregnancy test within 7 days before the index procedure, or lactating, or intends to become pregnant during the study
* Life expectancy of less than 24 months due to other medical conditions
* Co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
* Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study
* Left main coronary artery disease (stenosis >50%), whether protected or unprotected
* Target lesion is ostial in location (within 3.0 mm of vessel origin)
* Target lesion and/or target vessel proximal to the target lesion is severely calcified by visual estimation
* Target lesion involves a bifurcation with a diseased (>50% stenotic) branch vessel >2.0 mm in diameter that requires intervention
* Target lesion is totally occluded Thrombolysis In MI (TIMI flow ≤1)
* Angiographic presence of probable or definite thrombus
* Target vessel will be pre-treated with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon or transluminal extraction catheter immediately prior to stent placement
* Prior coronary intervention using brachytherapy to any segment of the target vessel
* The target vessel has had prior drug-eluting stent placement to vessel segment (or branch) proximal to intended target lesion site
* Angiographic restenosis of any segment of the target vessel that has undergone prior percutaneous coronary intervention
* Angiographic evidence of atherosclerotic disease with > 50% diameter stenosis (by visual estimate) proximal or distal to the target lesion (applies to the major epicardial portion of the target vessel and contiguous vessel segment if the target lesion is located in a branch vessel)
* Prior surgical revascularization of the target vessel with patent graft (saphenous vein graft or arterial conduit)
* Target lesion lies within 10 mm of prior surgical anastomosis site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Device Success | At procedure or hospital discharge

SECONDARY OUTCOMES:
Lesion success | 30 days, 6 months and 12 months
Procedure success | 30 days, 6 months and 12 months
Acute Device Performance | Index procedure
In hospital, 30-day, 6-month, 12-month MACE | 30-day, 6-month, 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Dubois, M.D., Principal Investigator — UH Gasthuisberg
Locations (1):
- UH Gasthuisberg, Leuven, Belgium